CLINICAL TRIAL: NCT06559904
Title: The Effect of Dıetary Interventıon in Adherence With The Medıterranean Dıet on Fatty Acid Parameters in Blood and Follicular Fluid Samples and Implantation Success in Women Undergoing Infertility Treatment
Brief Title: The Effect of the Mediterranean Diet on Fatty Acids in Biological Fluids of Women Undergoing Infertility Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Collaborators: Gazi University (Other)
Responsible Party: Principal Investigator, Özge CEMALİ, Res. Ass. Dr., Trakya University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 47/2020-06
Record Dates: First submitted 2024-08-09; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Women Diagnosed With Infertility
Keywords: Fatty acids, Folicular Fluid, Implantation, Infertility, Mediterranean Diet, Ratio of ω6/ω3fatty acid
MeSH Terms: conditions — Infertility | interventions — Diet, Mediterranean

STUDY DESIGN:
Intervention Model Description: First, the intervention group was created in the study and the study was completed, then the control group was studied. 5 interviews were conducted with the women in the intervention group and the average time between the first and last interviews was 15.03±1.59 weeks. 2 interviews were conducted with the women included in the control group and the time between these interviews was 1.41±0.53 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mediterranean diet (Other): Mediterranean diet was applied to this group according to the needs of the individuals. The explanation was made through the Mediterranean diet training document and sample menu prepared by the researcher. The individuals were asked to apply this diet for 12 weeks. The individuals' compliance with the diet was evaluated with food consumption records in 4-week periods. Blood samples were taken from the individuals at the beginning of the treatment as biological material and at the end, blood samples and follicle fluid samples were collected according to the adjuvant treatment. Fatty acid analyses were performed with gas chromatography.
  Interventions: Other: Mediterranean diet
- Control group (No Intervention): This group did not receive any intervention. Food consumption records, blood samples and follicular fluid samples were taken only once from individuals who came for IVF treatment.

INTERVENTIONS:
Other: Mediterranean diet — The 'Mediterranean Diet Education Document', prepared by the researcher, which includes general information about the characteristics of the Mediterranean diet and the portion sizes that should be followed daily and weekly, and information on how often, how much and when to consume food groups, was provided as a diet education, and information was provided on how to record three-day food consumption.
  A nutrition education compatible with the Mediterranean diet, organized by the researcher according to the individual's daily needs, was provided and a sample menu was explained to the individual face to face.
  Arms: Mediterranean diet

SUMMARY:
The aim of this study was to examine the effect of the Mediterranean diet, which is accepted as one of the adequate and balanced nutrition models today, as well as serum and follicular fluid fatty acid profile and implantation success in women with an age range of 19-40 (years) before infertility treatment. The study was conducted as a prospective and case-control study with a total of 32 volunteer women, 16 in the intervention group and 16 in the control group, who applied to Gazi University Hospital between February 2021 and February 2022.

ELIGIBILITY:
Inclusion Criteria:

Women diagnosed with infertility Women between the ages of 19-40 Women with BMI <30 kg/m² women undergoing assisted reproductive treatment in which updated oocytes and semen be used Women undergoing assisted reproductive treatment (ART), IUI or one of the first 3 IVF/ICSI treatments (number of ART treatments ≤ 3)

Exclusion Criteria:

Women diagnosed with chronic diseases other than infertility Women who smoke and drink alcohol Women on ART who will use frozen eggs or semen Women with BMI >30 kg/m2 at the first measurement Women experiencing communication breakdown/timeout, becoming pregnant, difficulty adhering to a diet program or ART while the intervention is ongoing

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2023-11-02 (Actual)

PRIMARY OUTCOMES:
first meeting | through study completion, an average of 1 year
  using the questionnaire form, applying anthropometric measurements, drawing blood samples, and recording food intake for three days
second meeting | through study completion, an average of 1 year
  An explanation of the individual Mediterranean diet
third and forth meeting | through study completion, an average of 1 year
  recording three-day food intake evaluate adherence to the Mediterranean diet using anthropometric measurements
fifth meeting | through study completion, an average of 1 year
  using the questionnaire form, applying anthropometric measurements, drawing blood samples, and recording food intake for three days, collecting follicular fluid samples

SECONDARY OUTCOMES:
analysis of blood and follicular fluid samples | through study completion, an average of 1 year
  Fatty acid analyses of the collected samples were performed by gas chromatography-flame ionization detector (GC-FID) at Gazi University Faculty of Pharmacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)